CLINICAL TRIAL: NCT03589261
Title: Hepatic Blood Flow Changes During Fluid Challenge Assessed by MRI in Volunteers Subjects: a Prospective Monocentric Study. PORTEAU Trial
Brief Title: Hepatic Blood Flow Changes During Fluid Challenge Assessed by MRI in Volunteers Subjects.
Acronym: PORTEAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2018_843_0006
Record Dates: First submitted 2018-07-03; First posted 2018-07-17 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Flow Changes
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI (magnetic resonance imaging) (Other): Hepatic blood flow baseline will be measured using MRI. Fluid challenge of 500 ml of NaCl 0.9% will be administered during 10 minutes. Before and After fluid challenge, MRI will be performed to compare flow changes.
  Interventions: Device: MRI (magnetic resonance imaging)

INTERVENTIONS:
Device: MRI (magnetic resonance imaging) — Fluid challenge will be performed with 500 ml of intra venous NaCl (0.9%). Hepatic blood flow measurement will be performed using MRI.
  Other Names: 500 ml of intra venous NaCl (0.9%).

SUMMARY:
Hepatic artery and portal flows are both regulated to assume the whole hepatic blood flow. Each counts for respectively 25% and 75%. That so-called "buffer response" assumes that when portal flow increases, hepatic artery flow decreases. During fluid challenge in intensive care unit, fluid challenge is often administered to improve hepatic perfusion. That observation is not demonstrated. The aim of the study is to test buffer response and portal flow during fluid challenge.

DETAILED DESCRIPTION:
Prospective monocentric study at Amiens Hospital University. 20 volunteers subjects will be include after providing informed consent. Fluid challenge will be performed with 500 ml of intra venous NaCl (0.9%). Hepatic blood flow measurement will be performed using MRI.

ELIGIBILITY:
Inclusion Criteria:

* Fasting for the last 12 hours.

Exclusion Criteria:

* Claustrophobia
* Any previous medical history disease;
* Any abdominal surgical disease
* Pregnancy or breastfeeding

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Portal blood flow measure before and after fluid challenge | Two hours: the difference in hepatic portal flow before and after a volume expansion of 500 ml NaCl 0.9%.
  Fluid challenge will be performed with 500 ml of intra venous NaCl (0.9%). Hepatic blood flow measurement will be performed using MRI (magnetic resonance imaging).

SECONDARY OUTCOMES:
Hepatic artery blood flow measure before and after fluid challenge | Two hours
  Hepatic artery blood flow measure before and after a volume expansion of 500 ml NaCl 0.9%.

OTHER OUTCOMES:
Flow ratio of portal flow on hepatic artery flow | Two hours
  Flow ratio of portal flow on hepatic artery flow before and after a volume expansion of 500 ml NaCl 0.9%.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

REFERENCES:
- [Result] Abou-Arab O, Beyls C, Moussa MD, Huette P, Beaudelot E, Guilbart M, De Broca B, Yzet T, Dupont H, Bouzerar R, Mahjoub Y. Portal Vein Pulsatility Index as a Potential Risk of Venous Congestion Assessed by Magnetic Resonance Imaging: A Prospective Study on Healthy Volunteers. Front Physiol. 2022 Apr 29;13:811286. doi: 10.3389/fphys.2022.811286. eCollection 2022. PMID 35574483